CLINICAL TRIAL: NCT00232999
Title: Efficacy/Safety Study of Nebulized IVX-0142, a Novel Antiallergic Drug, in Mild Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: AllerGen NCE Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IXR-201-04-142
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: Allergic asthma; Allergen challenge; Bronchial hyperresponsiveness
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Nebulized IVX-0142

SUMMARY:
This study is designed to evaluate the effectiveness of nebulized IVX-0142, a novel anti-allergic drug, to inhibit allergen-induced airway narrowing in patients with allergic asthma and the related increased sensitivity of the airways to other substances, as well as to investigate a possible anti-inflammatory effect of the drug in the airways.

ELIGIBILITY:
Inclusion Criteria:

* Mild stable allergic asthma
* Positive skin-prick test to at least one common aeroallergen
* Positive methacholine challenge
* Positive allergen-induced early- and late-phase airway bronchoconstriction
* General good health

Exclusion Criteria:

* Lung diseases other than mild allergic asthma
* History or symptoms of cardiovascular disease, significant neurologic disease, and/or clinically significant autoimmune disease
* Chronic use of asthma medications other than short or intermediate beta-agonists or ipratropium
* Use of tobacco products within one year starting study or smoking history >10 pack years
* If female, pregnant or lactating or have positive pregnancy test at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2005-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Serial lung function tests measured up to 7 hours post-allergen challenge to assess effects on early- and late-phase asthmatic reactions

SECONDARY OUTCOMES:
Methacholine PC20 pre- and post-allergen challenge
Anti-inflammatory activity in airways

CONTACTS AND LOCATIONS:
Overall Officials: Paul M O'Byrne, MD, Principal Investigator — McMaster University and AllerGen NCE
Locations (3):
- Canada (3):
  - Department of Medicine, McMaster University, Hamilton, Ontario
  - Centre de cardiology et de pneumologie de l'Universite Laval, Sainte-Foy (Quebec City), Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Duong M, Cockcroft D, Boulet LP, Ahmed T, Iverson H, Atkinson DC, Stahl EG, Watson R, Davis B, Milot J, Gauvreau GM, O'Byrne PM. The effect of IVX-0142, a heparin-derived hypersulfated disaccharide, on the allergic airway responses in asthma. Allergy. 2008 Sep;63(9):1195-201. doi: 10.1111/j.1398-9995.2008.01707.x. PMID 18699936